CLINICAL TRIAL: NCT06393114
Title: Impacts of Fermented Plant-based Products High in Protein and Fibre on Gut Microbiota and Health: a Randomized, Controlled, Cross-over Trial
Brief Title: Impacts of Fermented Oat-based Product on Gut Microbiota and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: University of Turku (Other); Umeå University (Other); ETH Zurich (Other); KU Leuven (Other)
Responsible Party: Principal Investigator, Marjukka Kolehmainen, Professor, University of Eastern Finland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HE 101060247
Record Dates: First submitted 2024-04-02; First posted 2024-05-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Syndrome
Keywords: Fermentation; Plant Proteins, Dietary; Inflammation Mediators; Gastrointestinal Microbiome; Tryptophan
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: During the run-in phase, participants consume their habitual diet. Subsequently, participants are randomized to incorporate one of the study products into their habitual diet for three weeks. The amount of the products to be consumed is 4-6 dl/day, with the precise amount being determined based on the participants' energy requirements. After the three-week diet period, participants will return to their habitual diet, followed by another three-week period during which they will consume the alternate intervention product. The overall duration of the study will be 12 weeks for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fermented product (Experimental): Participants will consume a fermented oat-based product daily for three weeks within their diet.
  Interventions: Other: Fermented oat-based product
- Unfermented product (Active Comparator): Participants will consume an unfermented oat-based product daily for three weeks within their diet.
  Interventions: Other: Unfermented oat-based product
- Habitual diet (No Intervention): Participants consume their habitual diet without any intervention products.

INTERVENTIONS:
Other: Fermented oat-based product — Participants will incorporate a novel fermented product into their habitual diet for three weeks. In addition, the consumption of dairy and plant-based dairy alternatives is restricted. Cereal product consumption, specifically bread and porridge, is slightly restricted to prevent gastrointestinal symptoms caused by the increased intake of dietary fibre. Participants will receive dietary guidance on how to follow the intervention diet, as well as potential supplement recommendations provided by the authorized nutritionist.
  Arms: Fermented product
Other: Unfermented oat-based product — Participants will incorporate a novel unfermented product into their habitual diet for three weeks. Dietary adjustments and other guidance are consistent with those described during the fermented product intervention.
  Arms: Unfermented product

SUMMARY:
This study aims to investigate the effects of consuming fermented oat-based products on gut and overall human health. It is a randomized, controlled, cross-over trial with a dietary intervention.

A total of 100 participants will be enrolled in this study and they will eat both fermented and unfermented oat-based products for three weeks. Participants will eat their habitual diet between the dietary intervention periods (wash-out).

During the study, participants' perceived health, inflammatory markers, glucose and lipid metabolism, tryptophan metabolites, gastrointestinal symptoms, and gut microbiota will be assessed.

DETAILED DESCRIPTION:
Plant-based protein sources, such as those derived from oats, are experiencing high demand due to their role in reducing reliance on animal products and promoting a more sustainable food system. Despite this, there is limited information available regarding the impact of components like fibre in plant-based foods on protein and other nutrients' metabolism.

Food fermentation emerges as a potential solution to enhance the absorption of plant-based protein and various nutrients in the small intestine. This is achieved by reducing antinutrients and facilitating the absorption process. Additionally, food fermentation has implications for the composition and metabolic activity of the gut microbiota, influencing metabolism, immune responses, intestinal function, and overall health. The metabolism of tryptophan in the gut, modulated by the gut microbiota and the production of various metabolites, may serve as a key link in these observed effects.

The fermentation of plant-based foods potentially enhances the beneficial health effects of these foods, and investigating this contributes to an increased understanding of the gut-mediated health effects of foods and the mechanisms behind them. This study will be part of a European research project HealthFerm.

Detailed objectives are to:

1. compare fermented and unfermented plant-based food products to blood lipid and glucose metabolism and gastrointestinal comfort as well as perceived and observed overall well-being.
2. study the effects of fermented and unfermented plant-based food consumption on the markers for gut permeability and inflammation.
3. study the difference in microbiota composition and diversity after consuming fermented and unfermented plant-based foods and its contribution to cardiometabolic outcomes.
4. study the difference in microbiota-related metabolites, especially tryptophan metabolites between fermented and unfermented plant-based foods.

A total of 100 participants will be enrolled in this randomized, controlled, cross-over trial, during which they will eat both fermented and unfermented oat-based products as part of their habitual diet. The study follows this sequence:

Weeks 1-3: Habitual diet Weeks 4-6: Dietary Intervention 1 Weeks 7-9: Habitual diet (wash-out) Weeks 10-12: Dietary Intervention 2

Blood, urinary and faecal samples, as well as food diaries and questionnaires, are collected at the end of each study period to assess participants' perceived health, inflammatory markers, glucose and lipid metabolism, tryptophan metabolites, gastrointestinal symptoms, and gut microbiota. In addition, participants' values and attitudes towards fermented foods are assessed. At the end of the study, participants will receive their laboratory results and dietary guidance for their habitual diet from a registered dietitian.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference >90 cm (women) or >100 cm (men) OR BMI 26-38 kg/m2
* One of the following:

  * raised blood pressure (systolic ≥ 130 mmHg and/or diastolic 85 mmHg)
  * raised fasting plasma glucose (≥ 5.6 mmol/l)
  * raised triglycerides (≥ 1.7 mmol/l)
  * raised total cholesterol (≥ 5 mmol/l)
  * raised LDL (≥ 3 mmol/l)
  * reduced HDL (women < 1.3 mmol/l, men 1.0 mmol/l)
* Use of cereal products and dairy products or their plant-based alternatives as a part of habitual diet
* Willingness to follow intervention diets for the whole study

Exclusion Criteria:

* Diagnosed chronic diseases and conditions which could hamper the adherence to the dietary intervention protocol, e.g., chronic liver, thyroid, kidney, or gastrointestinal diseases
* Pregnancy and lactation
* Gluten-free or vegan diet
* Recent use of antibiotics (within 3 months)
* Gastrointestinal surgery (within 6 months)
* Alcohol abuse (AUDIT ≥ 15 p and measures of liver function)
* regular smoking or use of snus

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker 1 | Weeks 3, 6, 9, and 12
  P-hs-CRP (mg/l)
Inflammatory marker 2 | Weeks 3, 6, 9, and 12
  IL-22
Inflammatory marker 3 | Weeks 3, 6, 9, and 12
  LBP (μg/ml)

SECONDARY OUTCOMES:
Changes in the composition gut microbiota | Weeks 3, 6, and 12
  Composition of gut microbiota will be analysed from faecal samples
Glucose metabolism | Weeks 3, 6, 9, and 12
  fP-Gluk and B-HbA1C (mmol/l)
Insulin response | Weeks 3, 6, 9, and 12
  fP-Insu (mU/l)
Lipid metabolism | Weeks 3, 6, 9, and 12
  fP-Kol, fP-Kol-HDL, fP-Kol-LDL, fP-Trigly, and fP-FFA (mmol/l)
Tryptophan metabolism | Weeks 3, 6, 9, and 12
  Tryptophan metabolites will be analysed with non-targeted metabolomics.
Self-reported overall health | Weeks 3, 6, 9, and 12
  Short Form-36 Health Survey (SF-36). Different sections are rated from 0 to 100 points, where higher scores mean better perceived health.
Self-reported mental health | Weeks 3, 6, 9, and 12
  General Health Questionnaire-12 (GHQ-12). The questionnaire is rated from 0 to 12 points, where higher score means greater psychological distress.
Self-reported gut health | Weeks 3, 6, 9, and 12
  Gastrointestinal Symptoms Rating Scale (GSRS)
Attitudes and values | Weeks 0 and 12
  Unvalidated questionnaire
Opinions about the study products | Weeks 6 and 12
  Unvalidated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marjukka Kolehmainen, Principal Investigator — Professor
Locations (1):
- University of Eastern Finland, Kuopio, Finland